CLINICAL TRIAL: NCT04435353
Title: Assessment of the Effectiveness of Vibroacoustic Therapy for Respiratory Failure Caused by COVID 19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Mukatova Irina, PhD. Professor of medicine. Head of deparment pulmonology, Astana Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AstanaMU
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Distress Syndrome; Hypoxemia
Keywords: Vibroacustic therapy; COVID19; Pneumonia
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia; COVID-19; Pneumonia

STUDY DESIGN:
Intervention Model Description: Prospective\retrospective study
Who Masked: Outcomes Assessor
Masking Description: Research involves single blinding (researcher statistician)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Time-day of respiratory fail (Active Comparator): Objective data
  Interventions: Device: VibroLUNG
- Oxygen status (Active Comparator): Facultative data
  Interventions: Device: VibroLUNG
- Oxugen support (Active Comparator): FiO2
  Interventions: Device: VibroLUNG
- Adverse outcomes (Active Comparator): Complication
  Interventions: Device: VibroLUNG

INTERVENTIONS:
Device: VibroLUNG — Lungs intensive therapy
  Other Names: Vibroacustic device

SUMMARY:
Vibroacoustic pulmonary therapy in patients with COVID19 is believed to have a positive effect on oxygen status and a decrease in the duration of respiratory failure

DETAILED DESCRIPTION:
This study aims to recruit the required number of patients for statistical identification of the effectiveness of vibroacoustic therapy in patients with COVID 19. Obligatory performance criteria will be presented by the duration of the course of respiratory failure and the duration of mechanical ventilation in the main and control groups. Optional performance criteria will be represented by oximetry values and standardization of laboratory parameters

ELIGIBILITY:
Inclusion Criteria:

1. adults
2. P/F less 300 torr
3. ARDS by Berlin convention
4. COVID 19 bilateral pneumonia

Exclusion Criteria:

1. children
2. acute brain stroke
3. acute coronary syndrome
4. pulmonary embolism
5. implanted pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Recovery respiratory fail | 5-7 days
  Regression of respiratory failure under the influence of vibroacoustic therapy

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - Mukatova Irina, Astana, Astana
  - Center of pulmonology Astana, Astana